CLINICAL TRIAL: NCT07112079
Title: Parental Perceptions of Antibiotic Use in Pediatric Dentistry: a Cross-sectional Study Using the PAPA Scale
Brief Title: Parental Views on Antibiotics in Dentistry
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2024/181
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Antibiotic; Oral Health Care; Parents; Pediatric Dentistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children (n=805): This cross-sectional study included a group of 805 children aged 3 to 14 years. Children's oral health was clinically evaluated using the DMFT (Decayed, Missing, and Filled Teeth) and PUFA (Pulpal involvement, Ulceration, Fistula, and Abscess) indices to provide an objective measure of dental health.
- Group 2: Parents (n=805): This cross-sectional study involved a cohort of 805 parents of children aged 3 to 14 years. The primary objective was to assess parental knowledge and attitudes towards antibiotic use. No interventions were implemented; instead, data were collected using a 45-item questionnaire based on the Parental Perceptions on Antibiotics (PAPA) scale. The PAPA scale evaluates various factors influencing parental decisions regarding antibiotic use, including knowledge, beliefs, behaviors, sources of information, adherence, and awareness of antibiotic resistance . The questionnaire was administered face-to-face to ensure accurate data collection and to facilitate clarification of any questions.

SUMMARY:
This study aims to assess parents' knowledge of antibiotic use and its relationship with their children's oral health.

DETAILED DESCRIPTION:
This study included 805 children (ages 3-14 years) and their parents. A face-to-face questionnaire with 45 items was used to assess parental knowledge and attitudes using the PAPA (Parental Perceptions on Antibiotics) scale. Children's oral health was clinically evaluated using DMFT (decayed, missing, and filled teeth) and PUFA (pulpal involvement, ulceration, fistula, and abscess) indices.

ELIGIBILITY:
Inclusion Criteria:

* Children whose parents were literate in Turkish, enabling reliable communication.
* Children whose parents had no communication impairments, ensuring accurate data collection.

Exclusion Criteria:

* Children who attended the clinic with a legal guardian or relative other than their parents.
* Children whose parents had inadequate health status preventing successful completion of the questionnaire.
* Children with any diagnosed mental illness.
* Children whose parents had any diagnosed mental illness.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Probability Sample
Enrollment: 1610 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Parental Knowledge and Beliefs on Antibiotic Use (Knowledge and Beliefs Subscale of the PAPA Scale) | 1 month
  Evaluation of parents' knowledge level and misbeliefs regarding antibiotic use: This score is obtained from the Knowledge and Beliefs subscale of the PAPA scale and measures the level of knowledge of parents on issues such as the necessity and appropriateness of antibiotics.
DMFT Index (Decayed, Missing, and Filled Teeth) Score | 1 month
  The DMFT index assesses the dental caries experience by counting the number of decayed, missing, and filled permanent teeth. Scores range from 0 to 28 (or 32 depending on dentition), where higher scores indicate worse dental health (more caries experience).
PUFA Index (Pulpal involvement, Ulceration, Fistula, and Abscess) Score | 1 month
  The PUFA index measures the clinical consequences of untreated dental caries, including pulpal involvement, ulceration, fistula, and abscess formation. Scores range from 0 to 4, where higher scores indicate more severe clinical complications due to untreated caries.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No